CLINICAL TRIAL: NCT04756973
Title: The Addition of Self-compassion Skills Training to a Behavioral Weight Loss Program Delivered Using Video Conferencing Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCIRB 20-001508
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard weight loss (Active Comparator): A 12 week small group weight loss intervention delivered via video teleconference technology.
  Interventions: Behavioral: Behavioral weight loss program
- Standard weight loss plus self-compassion skills training (Experimental): A 12 week small group weight loss intervention delivered via video teleconference technology.
  Interventions: Behavioral: Behavioral weight loss program

INTERVENTIONS:
Behavioral: Behavioral weight loss program — A 12 week small group weight loss program delivered via teleconference video technology

SUMMARY:
The current study examined the efficacy, feasibility, and acceptability of: 1) adding self-compassion (SC) skills training to a standard behavioral weight loss program (BWLP), and 2) utilizing video conferencing software to deliver small group, weekly, weight loss classes.

DETAILED DESCRIPTION:
Object: The current study examined the efficacy, feasibility, and acceptability of: 1) adding self-compassion (SC) skills training to a standard behavioral weight loss program (BWLP), and 2) utilizing video conferencing software to deliver small group, weekly, weight loss classes.

Method: The BWLP program utilized Webex video conferencing software to deliver a 12-week, interactive, small group, weekly weight loss intervention. Participants were randomized to a standard BWLP or a standard behavioral weight loss program augmented with self-compassion skills training (BWLP+SC).

ELIGIBILITY:
Inclusion Criteria:

* 18 or older, at a BMI of 27 kg/m2 or greater, and available to attend weekly online groups

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
weight loss | 12 weeks
  Weight in kilograms
height | baseline
  meters

SECONDARY OUTCOMES:
Self-compassion | 12 weeks
  Change in self-compassion scale score from pre to post
Eating Behaviors | 12 weeks
  Change in eating behaviors scale from pre to post

CONTACTS AND LOCATIONS:
Overall Officials: Robert Carels, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No